CLINICAL TRIAL: NCT06759298
Title: The Effects of Methylphenidate on Symptomatology in Individuals With Borderline Personality Disorder
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Osama Ibrahim Younes, lecturer of psychiatry, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: methylphenidate in borderline
Record Dates: First submitted 2024-12-10; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Borderline Personality Disorder
Keywords: methylphenidate
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Methylphenidate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Concerta Group (Active Comparator): Participants will receive a starting dose of Concerta (18 mg/day), which may be titrated based on clinical response and tolerance, up to a maximum of 54 mg/day. tablet form once daily for 3 months
  Interventions: Drug: methylphenidate
- Placebo Group (Placebo Comparator): Participants in the placebo group will receive a matched placebo tablet
  Interventions: Drug: matched placebo tablet

INTERVENTIONS:
Drug: methylphenidate — patient group will recieve methylphenidate
  Other Names: Concerta
  Arms: Concerta Group
Drug: matched placebo tablet — placebo gtoup will recieve matched placebo tablet
  Arms: Placebo Group

SUMMARY:
This study aims to investigate the effects of methylphenidate on symptomatology in individuals with borderline personality disorder. Specifically, it will evaluate whether Concerta is effective in reducing impulsivity, mood instability, and inattention among patients with BPD. Additionally, the study will assess Concerta's safety profile in this population to determine its potential as a supportive pharmacological option in BPD management.

DETAILED DESCRIPTION:
Borderline personality disorder (BPD) is a complex mental health condition characterized by pervasive instability in mood, self-image, interpersonal relationships, and behavior.

Individuals with BPD often experience intense episodes of anger, depression, and anxiety, which can lead to impulsive behaviors, self-harm, and strained social relationships. These symptoms significantly impair daily functioning and quality of life(American Psychiatric Association, 2013). creating a substantial burden on individuals and healthcare systems(Lieb et al., 2004).

. While psychotherapy remains the primary treatment for BPD, pharmacological interventions are often utilized to address specific symptoms, such as mood instability, impulsivity, and inattention.

Traditional medications like antidepressants, antipsychotics, and mood stabilizers have shown varying levels of efficacy in treating BPD, but no medication is currently approved specifically for BPD treatment(Chapman, 2019).. As a result, there is a growing interest in exploring alternative pharmacological options that may alleviate specific symptom clusters within BPD (Fleischhaker et al., 2011).

methylphenidate, a long-acting formulation of methylphenidate commonly prescribed for attention-deficit/hyperactivity disorder (ADHD), has shown promising effects on attention, impulsivity, and mood regulation(Hirsch & Hauschild, 2019).

These effects suggest it may be beneficial in managing certain BPD symptoms, particularly impulsivity and mood dysregulation. Preliminary studies have indicated that stimulant medications like methylphenidate may help some individuals with BPD improve focus and control impulsive behaviors, but comprehensive research on methylphenidate's efficacy and safety in this population remains limited(Wilens, Morrison, & Prince, 2011).

ELIGIBILITY:
Inclusion Criteria:

* • Individuals aged 18-50 years.

  * Diagnosed with borderline personality disorder as confirmed by a structured clinical interview.
  * Experiencing at least moderate levels of impulsivity and mood instability.
  * Not currently receiving stimulant medication or any pharmacotherapy specifically contraindicated with methylphenidate.
  * Capable of providing informed consent.

Exclusion Criteria:

* • Diagnosed with ADHD or other neurodevelopmental disorders where Concerta is typically prescribed.

  * Severe co-morbid psychiatric disorders (e.g., schizophrenia, bipolar disorder) or substance use disorder.
  * Known hypersensitivity to methylphenidate or other stimulant medications.
  * Pregnant or lactating women.
  * Individuals currently undergoing intensive psychotherapy or those unwilling to discontinue existing psychotropic medications that may interact with Concerta.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-03-25 (Estimated)

PRIMARY OUTCOMES:
Reduction in impulsivity and mood instability as measured by Barratt Impulsiveness Scale-11 (Revised) | 3 months
  Reduction in impulsivity and mood instability in borderline as measured by Barratt Impulsiveness Scale-11 (Revised)
reduction of depression symptoms in borderline personality as meassured by as measured by Barratt Impulsiveness Scale-11 (Revised) | 3 months
  reduction of depression symptoms in borderline personality as meassured by as measured by Barratt Impulsiveness Scale-11 (Revised)
Reduction in Perceived Stress in borderline as meassured by Perceived Stress Scale AScale | 3 months
  Reduction in Perceived Stress in borderline as meassured by Perceived Stress Scale

REFERENCES:
- [Background] Lieb K, Zanarini MC, Schmahl C, Linehan MM, Bohus M. Borderline personality disorder. Lancet. 2004 Jul 31-Aug 6;364(9432):453-61. doi: 10.1016/S0140-6736(04)16770-6. PMID 15288745